CLINICAL TRIAL: NCT00285506
Title: The Effect of Low-Osmolar and Iso-Osmolar Contrast Media on Erythrocytes in Healthy Volunteers.
Brief Title: The Effect of Contrast Media on Erythrocytes in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: GE Healthcare (Industry)
Other Study IDs: HR 15813
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2006-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of the study is to test the effect that contrast media (dye) has on cellular integrity (structure)

DETAILED DESCRIPTION:
The influence of several radiological contrast media on erythrocyte morphology and function has been investigated in the past (1). However, published data is sparse and does not include the assessment of iso-osmolar agents as compared to low-osmolar agents.

In addition, the effect of the injection of contrast media at higher temperatures (i.e. > room or body temperature), which may be beneficial for the rapid injection of more viscous contrast media at multi detector-row CT angiography, has never been evaluated.

We intend to assess the hypothesis, that iso-osmolar contrast media (i.e. Visipaque) exerts less effect on erythrocyte morphology and function as compared to low-osmolar agents.

In addition, we intend to identify the upper temperature limit, at which contrast media can be injected, without affecting erythrocyte integrity.

Subjects will have up tp 400 mLs (approximately 26 tablespoons) of blood drawn. The blood will be kept at body temperature in a petri dish or similar container and exposed to contrast media (dye).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years old
* Subjects must be at least 110lbs and

Exclusion Criteria:

* Subjects may not be pregnant
* Subjects must not possess any medical conditions that would preclude them from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: U. Joseph Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States